CLINICAL TRIAL: NCT04449042
Title: Pediatric Airway Management Complications During the COVID-19 Pandemic. An International, Multicenter, Observational Registry: The PAWS-COVID-19 (Pediatric AirWay complicationS COVID-19) Registry
Brief Title: The PAWS-COVID-19 (Pediatric AirWay complicationS COVID-19) Registry
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: Children's Hospital of Philadelphia (Other); Children's Hospital Colorado (Other); Istituto Giannina Gaslini (Other); The Hospital for Sick Children (Other); Perth Children's Hospital of Western Austrailia (Unknown); Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Mary Lyn Stein, Assistant in Perioperative Anesthesia, Boston Children's Hospital
Other Study IDs: IRB-P00035427
Record Dates: First submitted 2020-06-22; First posted 2020-06-26 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Airway Management; COVID19
Keywords: COVID19 pediatric; intubation; anesthesia
MeSH Terms: conditions — COVID-19 | interventions — Anesthesia, General

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- COVID19 positive: a recently performed test which is positive for coronavirus infection
  Interventions: Procedure: airway management during sedation or general anesthesia
- COVID19 negative: a recently performed test which is negative for coronavirus infection
  Interventions: Procedure: airway management during sedation or general anesthesia
- COVID19 presumed positive: patients who do not have testing or who have negative testing but whose symptoms, history, physical exam, laboratory and imaging findings are consistent with infection with COVID19 and are treated as positive
  Interventions: Procedure: airway management during sedation or general anesthesia
- COVID19 presumed negative: patients who do not have testing, but based on symptoms, history, physical exam, laboratory and imaging findings are deemed to be low risk for COVID19 infection and are treated as negative
  Interventions: Procedure: airway management during sedation or general anesthesia

INTERVENTIONS:
Procedure: airway management during sedation or general anesthesia — airway management in children receiving sedation or general anesthesia for an elective, emergency, or urgent diagnostic or surgical procedure

SUMMARY:
The COVID-19 pandemic has disrupted anesthesia care all over the world. There remains very little data on current practice patterns and patient outcomes, particularly in anesthetized children. This is a prospective observational, multi-center study to investigate airway management related outcomes in children undergoing anesthesia during this pandemic. The investigators will compare the incidence of complications (particularly hypoxemia) in patients with COVID-19 to those who are COVID-19 negative during airway management.

PAWS COVID-19 Registry https://is.gd/PEDICOVID19

Registration link https://is.gd/researchrequest

ELIGIBILITY:
Inclusion Criteria:

* Undergoing an inpatient or outpatient procedure under general anesthesia with or without regional analgesia
* Undergoing a diagnostic procedure under sedation or general anesthesia
* Undergoing an urgent or emergent procedure performed during and outside of the regular operating room schedule hours.

Exclusion Criteria:

* Age > 18 years.
* Children admitted to the operating room already intubated
* Children who require tracheal intubation for life-threatening conditions in the emergency department, intensive care, or hospital ward.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population will include all children (from birth to 18yrs) receiving sedation or general anesthesia for an elective, emergency, or urgent diagnostic or surgical procedure. Each institution will collect de-identified data on all children under anesthetic care for a two week period. In addition, data collection for all children who are positive or presumed positive for COVID19 receiving anesthetic care will be collected outside of the two week period until study completion.
Sampling Method: Non-Probability Sample
Enrollment: 14835 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
airway complications | throughout duration of anesthetic
  incidence of complications (particularly hypoxemia) in patients with COVID-19 to those who are COVID-19 negative during airway management

SECONDARY OUTCOMES:
airway device | throughout duration of anesthetic
  type of device inserted for airway control
PPE | throughout duration of anesthetic
  the type of PPE used by anesthetists and assistants during airway management
First pass success | during induction and intubation
  compare the first attempt success rate of tracheal intubation in patients with the disease to those without the disease
induction techniques | during induction of anesthesia
  variability in practice for induction of anesthesia
failed intubation | during induction of anesthesia
  determine the Incidence of failed intubation
complication risk factors | during anesthetic management
  determine risk factors related to complications (PPE type, Location, Age, Baseline Saturation, Induction technique, clinician type)

CONTACTS AND LOCATIONS:
Overall Officials: John E Fiadjoe, MD, Study Chair — Children's Hospital of Philadelphia; Melissa Brooks Peterson, MD, Principal Investigator — Colorado Children's Hospital
Locations (1):
- Boston Children's Hopsital, Boston, Massachusetts, United States